CLINICAL TRIAL: NCT00275639
Title: A Randomized, Double-blinded, Placebo-controlled Study of Angiotensin II Receptor Blockade to Prevent Renal Dysfunction Following Liver Transplantation.
Brief Title: The Effects of Angiotensin II Receptor Blockade on Kidney Function and Scarring After Liver Transplant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2085-04
Record Dates: First submitted 2006-01-10; First posted 2006-01-12 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Liver Transplant Recipients
MeSH Terms: interventions — Losartan

INTERVENTIONS:
Drug: Cozaar

SUMMARY:
This research study is being done to study the effects, both good and bad, of calcineurin inhibitors and the drug Cozaar (losartan), on kidney function and kidney scarring following a liver transplant.

DETAILED DESCRIPTION:
This study is a double-blinded, placebo controlled trial to help determine the pathogenesis of chronic renal dysfunction in patients undergoing liver transplantation. It will examine the renal function and renal morphology in patients on calcineurin inhibitors and the effects of Cozaar (losartan) following liver transplantation. Participants will have blood, urine and iothalamate clearance test, to look at kidney function prior to transplant. At the time of transplant, kidney biopsies will be performed in the operating room under anesthesia. Participants will be in the study for one year. At three weeks following liver transplant, participants will be randomly assigned to receive either a placebo (inactive drug) or the study drug (losartan). The participant will need to continue to return to the clinic at the normal scheduled intervals. During these times blood and urine tests will be done. A kidney biopsy will be performed at the yearly exam and study pills will be stopped. The researchers will continue to follow participant's creatine measurements for the next 10 years.

ELIGIBILITY:
Participants who will be undergoing a liver transplant and are between the ages of 18 to 70 years of age.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2004-12; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Development of renal dysfunction (measured by iothalamate clearance).

CONTACTS AND LOCATIONS:
Overall Officials: K.V. Narayanan Menon, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States